CLINICAL TRIAL: NCT02134301
Title: An Open Label, Dose-finding, Pharmacokinetics, Safety, and Tolerability Study of Oritavancin Single Dose Infusion in Pediatric Subjects Less Than 18 Years of Age With Suspected or Confirmed Bacterial Infections
Brief Title: Open Label, Dose-finding, Pharmacokinetics, Safety and Tolerability Study of Oritavancin in Pediatric Participants With Suspected or Confirmed Bacterial Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-ORI-11-01; 2013-005415-26 (EudraCT Number)
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Gram-positive Bacterial Infections
Keywords: Oritavancin; Pediatrics; Gram-positive; Bacterial Infection; Confirmed; Suspected
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Bacterial Infections | interventions — oritavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oritavancin (Experimental): Single-dose IV Oritavancin Diphosphate
  Interventions: Drug: Oritavancin

INTERVENTIONS:
Drug: Oritavancin

SUMMARY:
The purpose of this Phase 1 trial is to evaluate the pharmacokinetics (PK), safety and tolerability of oritavancin in participants <18 years old with a confirmed or suspected bacterial infection.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, PK, safety and tolerability study of oritavancin in pediatric participants (<18 years of age) with suspected or diagnosed Gram-positive bacterial infections or pediatric participants requiring peri-operative prophylactic antibiotics. Approximately 54 participants will be enrolled at 5-10 United States centers. This study will include 5 age cohorts and participants will be entered in a stepwise approach starting with the older age cohort (12 to <18 years). The starting dose will be intravenous (IV) oritavancin 15 milligrams/kilogram. The safety, tolerability and PK data will be reviewed at the completion of each cohort to ensure safety and determine the appropriate dose for the next age cohort. At least 8 participants will be enrolled in each cohort except for the birth to <3 month age cohort which will have at least 16 participants enrolled. Three PK samples will be collected over 14 days. The safety follow-up will complete with a 60-day phone call to the caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Males and females <18 years of age.
* Neonates must be at least 34 weeks post-conception age.
* Parent or legal guardian has given informed consent, as appropriate; and pediatric participant has given verbal assent where appropriate.
* Suspected or diagnosed Gram-positive bacterial infection for which the participant is receiving standard antibiotic therapy; or peri-operative prophylactic use of antibiotics.
* Intravenous access to administer study drug.
* The participant will be observed in the emergency room or hospital for at least 1 hour after the study drug infusion is completed.

Exclusion Criteria:

* Septic shock or acute haemodynamic instability.
* History of immune-related hypersensitivity reaction to glycopeptides (such as vancomycin, dalbavancin, televancin, or teicoplanin) or any of their excipients.
* Participants who have taken vancomycin, telavancin, teicoplanin or other glycopeptide within 24 hours of screening or who are anticipated to need these drugs within 48 hours after administration of study drug. Participants who have taken dalbavancin are excluded if taken within the previous 2 weeks or who are anticipated to need dalbavancin within 48 hours after administration of study drug.
* Females who are of childbearing potential and unwilling to practice abstinence or use at least two methods of contraception or female participants of childbearing who are lactating or have a positive pregnancy test result at screening.
* Males who are unwilling to practice abstinence or use an acceptable method of birth control during the entire study period.
* Any surgical or medical condition which, in the opinion of the investigator, would put the participant at increased risk or is likely to interfere with study procedures or PK of the study drug.
* Participants whom the investigator considers unlikely to adhere to the protocol, comply with study drug administration, or complete the clinical study.
* Treatment with investigational medicinal product or investigational device within 30 days (or 5 times the half-life of the investigational medicine, whichever is longer) before enrollment and for the duration of the study.
* Any clinically significant disease or condition affecting a major organ system, including but not limited to gastrointestinal, renal, hepatic, endocrinologic, broncho-pulmonary, neurological, metabolic or cardiovascular disease.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2014-05; Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter (Area under the plasma concentration time-curve [AUC]) | 336 hours post infusion start time for Cohorts 1-4 and 168 hours for Cohort 5
  PK parameters (AUC)

SECONDARY OUTCOMES:
Pharmacokinetic Parameters | 336 hours post infusion start time for Cohorts 1-4 and 168 hours for Cohort 5
  PK parameters (Cmax, half-life, tmax, volume of distribution and clearance)
Safety Endpoint | Up to Day 60 post-dose
  Safety of oritavancin assessed according to clinical laboratory parameters, and adverse events (AEs) and serious adverse events (SAEs) up to 60 days following termination of the study drug infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Melinta Therapeutics, Inc.
Locations (8):
- United States (8):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital, San Diego, California
  - UCLA Harbor Medical Center, Torrance, California
  - Univ of Louisville, Norton Children's Research Institute, Louisville, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Toledo Children's Hospital, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: Undecided